CLINICAL TRIAL: NCT04440696
Title: To Evaluate the Tolerance, pd, and pk of Lanthanum Polystyrene-sulfonate Powder in a Phase Ib/ IIa Clinical Trial in Patients With ESRD-HD Hyperphosphatemia With Multi-center, Multi-dose, Give the Drug Multiple Time
Brief Title: To Evaluate the Patient Tolerance, Pharmacodynamics and Pharmacokinetics of Lanthanum Polystyrene Sulfonate Powder
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grand Life Science (Liaoning) Co., Ltd. (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JBL-2019-001
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1:dose 1.5g (Experimental): There were 12 subjects in the group, 8 of whom took lanthanum polystyrene sulfonate powder, 2 took placebo, and 2 took positive control drug （lanthanum carbonate）
  Interventions: Drug: Lanthanum Polystyrene Sulphonate Powder; Drug: Lanthanum Carbonate 500 MG; Drug: Placebo
- group 2:dose 3g (Experimental): There were 12 subjects in the group, 8 of whom took lanthanum polystyrene sulfonate powder, 2 took placebo, and 2 took positive control drug （lanthanum carbonate）
  Interventions: Drug: Lanthanum Polystyrene Sulphonate Powder; Drug: Lanthanum Carbonate 500 MG; Drug: Placebo
- group 3:dose 4.5g (Experimental): There were 12 subjects in the group, 8 of whom took lanthanum polystyrene sulfonate powder, 2 took placebo, and 2 took positive control drug （lanthanum carbonate）
  Interventions: Drug: Lanthanum Polystyrene Sulphonate Powder; Drug: Lanthanum Carbonate 500 MG; Drug: Placebo
- group 4:dose 6g (Experimental): There were 12 subjects in the group, 8 of whom took lanthanum polystyrene sulfonate powder, 2 took placebo, and 2 took positive control drug （lanthanum carbonate）
  Interventions: Drug: Lanthanum Polystyrene Sulphonate Powder; Drug: Lanthanum Carbonate 500 MG; Drug: Placebo

INTERVENTIONS:
Drug: Lanthanum Polystyrene Sulphonate Powder — D1 was administered once; D2-D12 was administered three times a day; D13 was administered once；
Drug: Lanthanum Carbonate 500 MG — D1 was administered once; D2-D12 was administered three times a day; D13 was administered once；
Drug: Placebo — D1 was administered once; D2-D12 was administered three times a day; D13 was administered once；

SUMMARY:
The aim of the study is:

To evaluate the tolerance of lanthanum polystyrene sulfonate powder in patients with end-stage renal disease (ESRD-HD) hyperphosphatemia with multiple doses and multiple doses； To evaluate the pharmacodynamics of lanthanum polystyrene sulfonate powder in hyperphosphatemia patients with end-stage renal disease on hemodialysis (ESRD-HD); To evaluate the pharmacokinetics of lanthanum polystyrene sulfonate powder in patients with end-stage renal disease (ESRD-HD) hyperphosphatemia after multi-dose and multiple administration.

ELIGIBILITY:
Inclusion Criteria(Only if all the criteria are met):

* 1) Sign the informed consent before the trial, and fully understand the test content, process and possible adverse reactions;
* 2) Able to complete the study according to the requirements of the experimental program, able to accept dietary management and unified diet during the trial;
* 3) Regular hemodialysis was performed three times a week in the 12 weeks before screening (the total number of weeks without three times a week for special reasons should not exceed 2 weeks), and the dialysis regimen was expected to remain unchanged during the trial;
* 4) The patient is receiving appropriate dialysis treatment, and the urea clearance index (KT /V) ≥1.2 (the KT /V value of the research center within one month before screening is valid, and the results of several measurements shall be subject to the latest measurement);
* 5) Subjects (including partners) are willing to voluntarily use effective contraceptive measures within 6 months from the screening to the last study drug administration, as detailed contraceptive measures are shown in Appendix 4;
* 6) Male and female subjects aged 18 to 65 years (including 18 and 65 years) with a body mass index (BMI) in the range of 18 to 35 kg/m2 (including the threshold);
* 7) In patients with end-stage renal disease hyperphosphatemia, fasting blood phosphorus ≥1.78mmol/L and ≤3.23mmol/L were measured at screening and admission.

Exclusion Criteria(If one of the exclusion criteria is satisfied, it is excluded):

* 1) A history of clinically significant drug allergy or atopic allergic disease (asthma, urticaria, eczema dermatitis) or known allergy to the experimental drug or similar drug;
* 2) Patients who had severe trauma or had undergone major surgery within 6 months prior to the trial, or who planned to undergo surgery during the study period were screened;
* 3) Blood loss > 450mL in the three months before screening;
* 4) Clinical, radiological or laboratory evidence of active tuberculosis (TB);
* 5) Previous kidney transplantation operations;
* 6) A history of drug use and/or alcohol abuse in the 3 months prior to screening (14 units of alcohol consumed per week: 1 unit = 285 mL beer, 25 mL spirits, or 100 mL wine);
* 7) Those who were receiving any vitamin D or calcium-like regimens at the time of screening and could not maintain a stable dose after admission (except those who were receiving a stable vitamin D or calcium-like regimens);
* 8) Have dysphagia or gastrointestinal history with any influence on drug absorption, including but not limited to intestinal obstruction, macrocolon, habitual constipation (stool frequency < 1 times per week), chronic diarrhea (stool frequency ≥4 times per day), gastroparesis with nausea or vomiting and other gastrointestinal disorders and gastrointestinal surgery;
* 9) suffer from any disease that increases the risk of gastrointestinal bleeding, such as acute erosive gastritis, acute hemorrhagic necrotizing enteritis, or active gastrointestinal ulcer;
* 10) For poorly controlled hypertension, the systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg should be measured at rest, and the patient should be rechecked at most twice for confirmation;
* 11) The history of acute coronary syndrome (such as myocardial infarction, unstable angina pectoris hospitalization), or percutaneous coronary intervention, or coronary artery bypass grafting in the previous 12 months was screened;Or had an arterial/venous thrombosis event, such as a cerebrovascular accident (including a history of stroke or transient ischemic attack), deep venous thrombosis and pulmonary embolism, within 12 months before screening;
* 12) Uncontrolled severe arrhythmias, such as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular response, or supraventricular tachycardia, that were not controlled by medication or other treatment in the 12 months prior to enrolment;
* 13) Unstable and serious diseases of the digestive system, respiratory system, mental nervous system, endocrine system, blood system, malignant tumor, etc., which are not suitable for the study as judged by the study doctor;
* 14) Screening patients with a history of acute or severe infection within the previous 1 month;
* 15) Take phosphorus-reducing drugs, such as lanthanum carbonate, calcium carbonate, calcium acetate, aluminum hydroxide, Sveram, etc., within 14 days before administration;Drugs that may affect lanthanum ion release, such as proton pump inhibitors, H2 receptor antagonists, etc.And drugs that interact with experimental drugs, such as ciprofloxacin hydrochloride, thyroxine, lithium, etc.;Drugs containing phosphoric acid components, such as oseltamivir phosphate, sitagliptin phosphate tablets, etc.
* 16) Those who have participated in any clinical trials of drugs or medical devices within one month before taking the study drug;
* 17) During screening, hemoglobin ≤90g/L and albumin ≤30g/L;
* 18) Hypercalcemia, blood calcium ≥2.52mmol/L;Hypocalcemia, blood calcium ≤1.80mmol/L (corrected blood calcium value: corrected blood calcium value mmol/L= measured calcium value mmol/L+0.02× (40g/L- measured serum albumin value g/L));
* 19) Severe hyperparathyroidism, parathyroid hormone (PTH) >1200pg/mL;
* 20) Female subjects with positive blood pregnancy results during the screening period or baseline period;
* 21) HIV antigen/antibody positive;Positive antibody to Treponema pallidum and positive serological test of non-Treponema pallidum (such as rapid plasma reaction test, toluidine red unheated serum test, etc.);
* 22) A history of heart failure as defined by the New York College of Cardiology (NYHA) as III-IV, or a left ventricular ejection fraction less than 40%;
* 23) Subjects who have other factors considered by the investigator to be unsuitable for participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood phosphate concentrations | At pre-defined intervals from initial dose through final study visit（Day -1 to Day 17）
Plasma lanthanum concentrations | At pre-defined intervals from initial dose through final study visit（Day -1 to Day 17）

SECONDARY OUTCOMES:
24h Urinary phosphate concentrations | At pre-defined intervals from initial dose through final study visit（Day 1 to Day 13）
Plasma PTH concentrations | At pre-defined intervals from initial dose through final study visit（Day 1 to Day 17）
Plasma calcium concentrations | At pre-defined intervals from initial dose through final study visit（Day 1 to Day 17）

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Ph.D, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No